CLINICAL TRIAL: NCT00083473
Title: A Pilot Study of Pivanex, a Histone Deacetylase Inhibitor, in Patients With Chronic Lymphocytic Leukemia
Brief Title: A Pilot Study of Pivanex in Patients With Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIV-801
Record Dates: First submitted 2004-05-24; First posted 2004-05-26 (Estimated); Last update posted 2005-08-30 (Estimated); Status verified 2005-08

CONDITIONS: Leukemia, Lymphocytic, Chronic; Lymphoma, Small Lymphocytic
Keywords: Leukemia Lymphocytic Chronic,; Pivanex,; Histone deacetylase inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell | interventions — pivalyloxymethyl butyrate

INTERVENTIONS:
Drug: Pivanex

SUMMARY:
This pilot study will assess the safety and efficacy of Pivanex alone in patients with chronic lymphocytic leukemia (CLL) who have relapsed or refractory disease after previous chemotherapy treatment. Pivanex is an investigational agent.

DETAILED DESCRIPTION:
Rationale: Chronic lymphocytic leukemia (CLL) is a disease characterized by the accumulation of mature lymphocytes. These CLL lymphocytes are blocked from undergoing terminal differentiation and apoptosis. Patients with CLL have limited options for therapy, especially after the failure of standard chemotherapy regimens. Histone deacetylase inhibitors (HDACs) comprise a new class of drugs being evaluated in the treatment of various malignancies. In vitro data suggest that HDAC inhibition leads to terminal B-cell differentiation and may therefore play a therapeutic role in the treatment of CLL. Pivanex (pivaloyloxymethyl butyrate) is an HDAC inhibitor that has been shown to induce apoptosis of CLL lymphocytes in vitro. In previous clinical trials, Pivanex has been well tolerated. The goal of this protocol is to determine the effects of Pivanex in patients with CLL.

Purpose: This open-label trial will determine the response rate of Pivanex in patients with CLL.

Objectives: (1) Determine the response rate of Pivanex in patients with relapsed CLL; (2) Determine time to disease progression in patients with relapsed CLL treated with Pivanex; and (3) Determine the safety profile of Pivanex in CLL.

Design: This is an open label, single arm, multiple dose, pilot study of patients with relapsed CLL. Patients will be treated with 2.5 g/m2 of Pivanex administered intravenously over 6 hours daily on Days 1 - 3. Treatment will be repeated every 21 days until disease progression or the patient is withdrawn from treatment for protocol-specified reasons.

Disease status will be assessed prior to every odd-numbered treatment cycle using response criteria based upon the Revised National Cancer Institute-sponsored Working Group Guidelines for CLL. Patients withdrawn due to disease progression will be followed for survival. Patients withdrawn from study for reasons other than disease progression will be followed for disease progression and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of CLL or small lymphocytic lymphoma (SLL) based upon the Revised NCI-sponsored Working Group guidelines for CLL;
* Relapsed or refractory disease after previous chemotherapy treatment;
* Age > 18 years;
* Adequate renal function with creatinine <= 1.5 mg/dL;
* Adequate liver function with alkaline phosphatase <= 2.5 X upper limit of normal, serum glutamic oxaloacetic transaminase (SGOT), and serum glutamic pyruvic transaminase (SGPT) <= 2.5 X upper limit of normal; and total bilirubin <= 2.0 X upper limit of normal;
* Adequate bone marrow function as determined by having platelets > 50,000/mm3 without transfusion in the preceding 2 weeks and an absolute neutrophil count (ANC) => 1,500 cells/mm3 without growth factor support; unless cytopenias due to marrow infiltration;
* Able to give informed consent;
* A minimum of 4 weeks must have elapsed from the completion of any previous treatment regimen, including radiation and biologic therapies (6 weeks if a prior nitrosourea or mitomycin C, 12 weeks if radioimmunotherapy) to treatment on Day 1 Cycle 1. Patients must have recovery from treatment-associated toxicity(ies);
* A predicted life expectancy of at least 6 months; and
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

* More than three systemic treatment regimens for CLL/SLL (excluding immunotherapies and biologic therapies);
* Concurrent malignancy that the patient has not been free of for at least 5 years, excluding curatively treated carcinoma-in-situ or non-melanoma skin cancer;
* Any pregnant or lactating females. Females of childbearing potential must have a negative pregnancy test and all male and female patients of reproductive potential must agree to use adequate birth control;
* Known HIV-positive patients;
* Any underlying medical conditions or circumstances that would contraindicate therapy with study treatment, affect compliance or impair evaluation of study endpoints;
* Receiving investigational agents within 4 weeks of the study treatment; and
* Known allergy to reagents in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2004-05; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Lymphoma and Myeloma; Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- See also: Click here for more information about study PIV-801 — http://www.titanpharm.com